CLINICAL TRIAL: NCT02756962
Title: Improving Risk Assessment of AML With a Precision Genomic Strategy to Assess Mutation Clearance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); American Society of Hematology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201606003
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cohort A: HiDAC (Experimental): * At the time of diagnostic bone marrow biopsy, samples will be clinically sequenced via ClinSeq
  * Patients who have clearance of their leukemia-associated mutations, defined as a LAM VAF <2.5% will be assigned to the high-dose cytarabine consolidation (HiDAC) arm.
  * HiDAC = Standard regimen of cytarabine 1.5 g/m^2 or 3 g/m^2 over 2-3 hours twice a day on Days 1, 3, & 5 of each 28 day cycle for 3-4 cycles. Can be replaced by Onureg with permission from PI.
  * For patients with the FLT3-ITD or a FLT3-TKD mutation, therapy with the FDA-approved FLT3 inhibitor midostaurin is permitted at the discretion of the treating physician.
  Interventions: Drug: Cytarabine; Procedure: Bone marrow aspiration; Procedure: Punch skin biopsy; Device: ClinSeq
- Cohort B: Investigator's choice (HiDAC, AlloSCT) (Experimental): * At the time of diagnostic bone marrow biopsy, samples will be clinically sequenced via ClinSeq
  * Patients who have persistent leukemia-associated mutations, defined as a LAM VAF ≥2.5% will be assigned to the investigator's choice arm.
  * Patients assigned to this arm may received either HiDAC or AlloSCT.
  * HiDAC = Standard regimen of cytarabine 1.5 g/m^2 or 3 g/m^2 over 2-3 hours twice a day on Days 1, 3, & 5 of each 28 day cycle for 3-4 cycles. Can be replaced by Onureg with permission from PI.
  * The source of stem cell product, donor selection, conditioning regimen, graft-versus-host-prophylaxis, and supportive care will be at the discretion of the treatment physician
  * For patients with the FLT3-ITD or a FLT3-TKD mutation, therapy with the FDA-approved FLT3 inhibitor midostaurin is permitted at the discretion of the treating physician.
  Interventions: Drug: Cytarabine; Procedure: Allogeneic stem cell transplant; Procedure: Bone marrow aspiration; Procedure: Punch skin biopsy; Device: ClinSeq

INTERVENTIONS:
Drug: Cytarabine
  Other Names: Ara-C; Cytosar-U; Tarabine-PFS; AraC
Procedure: Allogeneic stem cell transplant
  Other Names: AlloSCT
  Arms: Cohort B: Investigator's choice (HiDAC, AlloSCT)
Procedure: Bone marrow aspiration — * Baseline
  * Approximately 30 days after cytotoxic induction therapy
  * End of treatment
Procedure: Punch skin biopsy — * The first will be obtained with the initial blood and bone marrow collections, whenever possible.
  * The second will be obtained at the time of re-biopsy to confirm remission.
Device: ClinSeq — Clinical Sequencing to determine clearance or persistence of leukemia-associate mutations performed at MGI CLIA lab

SUMMARY:
The investigators will prospectively determine whether the relapse-free and overall survival in patients who have cleared their leukemia-associated mutations treated with standard consolidation chemotherapy is superior to what is expected based on historical controls. The investigators will also prospectively determine the relapse-free and overall survival of patients who have not cleared their mutations. Because the relapse rate of patients with persistent mutations is expected to be high, treatment with either standard of care consolidation therapy alone or alloSCT will be permitted, at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years.
* Considered to be suitable intensive (cytotoxic) induction candidates.
* Has previously untreated, de novo, non-M3 AML with intermediate-risk disease (Intermediate-I or Intermediate-II) as defined by ELN criteria OR normal cytogenetics with mutated NPM1 without FLT3-ITD. Monoallelic CEBPA mutations are not considered favorable risk and are therefore eligible.
* Has undergone cytotoxic induction therapy
* In a morphologic complete remission with incomplete blood count recovery, or morphologic complete remission post-induction after no more than 2 induction cycles as defined by revised IWG criteria
* Patients at Washington University must be enrolled in HRPO# 201011766 ("Tissue Acquisition for Analysis of Genetic Progression Factors in Hematologic Diseases").This is not a requirement for secondary sites. However, secondary sites must provide informed consent forms that document that permission for whole genome, whole exome, and/or genome wide sequencing, and data sharing among institutions, was obtained. Because we will be also be sequencing non-diseased (normal) tissue, the informed consent forms must explicitly ask if patients wish to be informed, (or in the case of their death, their next-of-kin) if a deleterious mutation is identified in their non-diseased tissue, as this may be heritable.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document.
* Willing to comply with the treatment assignment:

  * Intent to proceed with HiDAC consolidation for LAM VAF <2.5%
  * Intent to proceed with either HiDAC consolidation or allogeneic stem cell transplantation, at the discretion of the treating physician, for LAM ≥2.5%

Exclusion Criteria:

* Diagnosis acute promyelocytic leukemia (APL) with t(15;17)(q22;q12); PML-RARA.
* Therapy-related AML (defined as occurrence of AML due to prior exposure to chemotherapy or radiation for malignancy).
* Secondary AML (defined as development of AML in patients with an antecedent hematological malignancy).
* Has a medical or psychosocial conditions that would prevent study compliance.
* Known seropositivity for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B vaccine are eligible.
* History of allergic reaction to compounds of similar chemical or biologic composition to cytarabine.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 3 days of signing consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival of Cohort A compared to intermediate risk historical control group | Up to 5 years
  * Relapse-free survival is the time from study enrollment (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) is required) until documented disease relapse, or death from any cause.
  * CR=Defined as morphologic leukemia-free state, defined as less than 5% blasts in aspirate with marrow spicules and a count of ≥200 nucleated cells and no blasts with Auer rods or any persistence of extramedullary disease. In addition, ANC >1000/μl and platelet count of ≥100,000/μl. Patient must be independent of transfusions. No duration requirement for this designation.
  * CRi=Defined as morphologic complete recovery with the exception of neutropenia <1000/μl or thrombocytopenia <100,000/μl.

SECONDARY OUTCOMES:
Overall survival (OS) of Cohort A compared intermediate risk historical control group | Up to 5 years
  Overall survival is the time from enrollment on study until death from any cause.
Relapse free survival (RFS) of Cohort B | Up to 5 years
  * Relapse-free survival is the time from study enrollment (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) is required) until documented disease relapse, or death from any cause.
  * CR=Defined as morphologic leukemia-free state, defined as less than 5% blasts in aspirate with marrow spicules and a count of ≥200 nucleated cells and no blasts with Auer rods or any persistence of extramedullary disease. In addition, ANC >1000/μl and platelet count of ≥100,000/μl. Patient must be independent of transfusions. No duration requirement for this designation.
  * CRi=Defined as morphologic complete recovery with the exception of neutropenia <1000/μl or thrombocytopenia <100,000/μl.
Overall survival (OS) of Cohort B | Up to 5 years
  Overall survival is the time from enrollment on study until death from any cause.
Compare relapse free survival of Cohort A to Cohort B | Up to 5 years
  * Relapse-free survival is the time from study enrollment (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) is required) until documented disease relapse, or death from any cause.
  * CR=Defined as morphologic leukemia-free state, defined as less than 5% blasts in aspirate with marrow spicules and a count of ≥200 nucleated cells and no blasts with Auer rods or any persistence of extramedullary disease. In addition, ANC >1000/μl and platelet count of ≥100,000/μl. Patient must be independent of transfusions. No duration requirement for this designation.
  * CRi=Defined as morphologic complete recovery with the exception of neutropenia <1000/μl or thrombocytopenia <100,000/μl.
Compare overall survival of Cohort A to Cohort B | Up to 5 years
  Overall survival is the time from enrollment on study until death from any cause.
Compare relapse free survival of Cohort A to Cohort B | 1 year
  * Relapse-free survival is the time from study enrollment (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) is required) until documented disease relapse, or death from any cause.
  * CR=Defined as morphologic leukemia-free state, defined as less than 5% blasts in aspirate with marrow spicules and a count of ≥200 nucleated cells and no blasts with Auer rods or any persistence of extramedullary disease. In addition, ANC >1000/μl and platelet count of ≥100,000/μl. Patient must be independent of transfusions. No duration requirement for this designation.
  * CRi=Defined as morphologic complete recovery with the exception of neutropenia <1000/μl or thrombocytopenia <100,000/μl.
Compare overall survival of Cohort A to Cohort B | 1 year
  Overall survival is the time from enrollment on study until death from any cause.
Relapse free survival of Cohort B patients who receive alloSCT | Up to 5 years
  * Relapse-free survival is the time from study enrollment (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) is required) until documented disease relapse, or death from any cause.
  * CR=Defined as morphologic leukemia-free state, defined as less than 5% blasts in aspirate with marrow spicules and a count of ≥200 nucleated cells and no blasts with Auer rods or any persistence of extramedullary disease. In addition, ANC >1000/μl and platelet count of ≥100,000/μl. Patient must be independent of transfusions. No duration requirement for this designation.
  * CRi=Defined as morphologic complete recovery with the exception of neutropenia <1000/μl or thrombocytopenia <100,000/μl.
Overall survival of Cohort B patients who receive alloSCT | Up to 5 years
  Overall survival is the time from enrollment on study until death from any cause.
Relapse free survival of Cohort B patients who do not receive alloSCT | Up to 5 years
  * Relapse-free survival is the time from study enrollment (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) is required) until documented disease relapse, or death from any cause.
  * CR=Defined as morphologic leukemia-free state, defined as less than 5% blasts in aspirate with marrow spicules and a count of ≥200 nucleated cells and no blasts with Auer rods or any persistence of extramedullary disease. In addition, ANC >1000/μl and platelet count of ≥100,000/μl. Patient must be independent of transfusions. No duration requirement for this designation.
  * CRi=Defined as morphologic complete recovery with the exception of neutropenia <1000/μl or thrombocytopenia <100,000/μl.
Overall survival of Cohort B patients who do not receive alloSCT | Up to 5 years
  Overall survival is the time from enrollment on study until death from any cause.
Relapse free survival of patients with a LAM VAF <1.0% treated in Cohort A compared to intermediate risk historical control group | Up to 5 years
  * LAM VAF = Leukemia Associated Mutations variant allele frequency
  * Relapse-free survival is the time from study enrollment (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) is required) until documented disease relapse, or death from any cause.
  * CR=Defined as morphologic leukemia-free state, defined as less than 5% blasts in aspirate with marrow spicules and a count of ≥200 nucleated cells and no blasts with Auer rods or any persistence of extramedullary disease. In addition, ANC >1000/μl and platelet count of ≥100,000/μl. Patient must be independent of transfusions. No duration requirement for this designation.
  * CRi=Defined as morphologic complete recovery with the exception of neutropenia <1000/μl or thrombocytopenia <100,000/μl.
Overall survival of patients with a LAM VAF <1.0% treated in Cohort A compared to intermediate risk historical control group | Up to 5 years
  --LAM VAF = Leukemia Associated Mutations variant allele frequency
  -Overall survival is the time from enrollment on study until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu